CLINICAL TRIAL: NCT02588586
Title: An Open Label, Phase 2 Study of the Safety and Antiretroviral Activity of 3BNC117 in HIV-Infected Individuals on Combination Antiretroviral Therapy
Brief Title: A Study of the Safety and Antiretroviral Activity of 3BNC117
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Bill and Melinda Gates Foundation (Other); Weill Medical College of Cornell University (Other); Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Marina Caskey, MD, Assistant Professor of Clinical Investigation, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCA-0866; 1U01AI118536-01 (NIH)
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: HIV-1 Infection
Keywords: HIV; 3BNC117; Broadly neutralizing antibody
MeSH Terms: interventions — 3BNC117 antibody; Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3BNC117 + ART Interruption (Experimental): Four intravenous infusions of 3BNC117 (30mg/kg) at weeks 0, 12, 24 and 27, and antiretroviral treatment interruption (ART)at week 24.
  Interventions: Drug: 3BNC117; Other: Antiretroviral Treatment Interruption

INTERVENTIONS:
Drug: 3BNC117 — 3BNC117 infusions
  Other Names: 3BNC117 antibody
Other: Antiretroviral Treatment Interruption — Antiretroviral therapy will be discontinued 2 days after the third 3BNC117 infusion, at week 24, and resumed at week 36.
  Other Names: Treatment Interruption

SUMMARY:
This study evaluates the effects of four infusions of 3BNC117 in preventing or delaying rebound of viral load during a brief treatment interruption of standard ART, and its safety during a brief analytical interruption of antiretroviral therapy.

DETAILED DESCRIPTION:
The proposed study is a Phase II, open label study to evaluate the safety, antiretroviral activity and pharmacokinetics of four infusions of 3BNC117 in HIV-infected individuals on combination ART and during a brief analytical treatment interruption (ATI).

Study participants will be administered four intravenous infusions of 3BNC117, administered at 30 mg/kg on day 0, week 12, week 24 and week 27. Antiretroviral therapy will be discontinued 2 days after the third 3BNC117 infusion (week 24), until week 36.

The ART regimen will be resumed at week 36 or sooner if plasma HIV-1 RNA level is ≥ 200 copies/ml, CD4+ T cell count drops < 350 cells/microliter, and results are confirmed upon repeat measurement during the next weekly scheduled visit. If plasma HIV-1 RNA level is ≥ 1,000 copies/ml, the participant will be asked to return for a repeat measurement prior to the next scheduled visit, and ART will be resumed if results are confirmed. ART will also be resumed early if the participant becomes pregnant or if otherwise clinically indicated. If ART is resumed before week 27, the fourth 3BNC117 infusion will not be administered.

Participants will be followed weekly during the analytical treatment interruption phase for safety assessments and for monitoring plasma HIV-1 RNA levels. CD4+ T cell counts will be monitored every 2 weeks during the analytical treatment interruption phase.

Participants may remain off antiretroviral therapy after week 36, with weekly viral load monitoring, if viral rebound does not occur by week 36.

All participants will be followed for a total of 60 weeks from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and signed.
* Males and females, age 18 to 65.
* HIV-1 infection confirmed by two independent methods.
* Plasma HIV-1 RNA < 50 copies/ml for at least 12 months while on combination ART and < 20 copies/ml at the screening visit. [Note: One or two viral blips of < 200 copies/mL prior to enrollment are permitted if preceded and followed by test results showing VL less than or equal to 50 copies/ml on the same ARV regimen.]
* CD4 cell count > 500 cells/microliter. CD4 cell count nadir > 200 cells/microliter.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use an effective method of contraception throughout the study period. Participants should also agree to use a male or female condom while off ART.
* Female study participants of reproductive potential are defined as pre-menopausal women who have not had a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Women are considered menopausal if they have not had a menses for at least 12 months and have a FSH of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.
* Acceptable forms of contraception must include one of the following: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, IUD, or hormone-based contraceptive.
* If on an NNRTI-based regimen willing to a switch for 4 weeks to a dolutegravir-based regimen.

Exclusion Criteria:

* Have a history of AIDS-defining illness within 1 year prior to enrollment.
* Have a history of resistance to two or more antiretroviral drug classes.
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Chronic hepatitis B or hepatitis C.
* Participant report, or chart history, of significant coronary artery disease, myocardial infarction, percutaneous coronary intervention with placement of cardiac stents.
* Participant report, or chart history, of diabetes type 1 or 2 and/or current use of insulin or oral hypoglycemic medications.
* Uncontrolled hypertension, as defined by a systolic blood pressure > 180 and/or diastolic blood pressure > 120, in the presence or absence of anti-hypertensive medications.
* Total cholesterol level > 240 mg/dl or LDL level > 190 mg/dl at screen.
* Known family history of myocardial infarction or stroke in a first-degree relative aged < 60 years.
* Any other clinically significant acute or chronic medical condition, such as autoimmune diseases, that in the opinion of the investigator would preclude participation.
* Current cigarette use in excess of 1 pack per day;
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count less than or equal to 1,000 cells/microliter
* Hemoglobin less than or equal to 10 g/dL
* Platelet count less than or equal to 125,000 cells/microliter
* ALT greater than or equal to 2.0 x ULN
* AST greater than or equal to 2.0 x ULN
* Total bilirubin greater than or equal to 1.5 ULN
* Creatinine greater than or equal to 1.1 x ULN
* Coagulation parameters greater than or equal to 1.5 x ULN.
* Current antiretroviral regimen includes maraviroc or enfuvirtide.
* Pregnancy or lactation.
* Any vaccination within 14 days prior to 3BNC117 administration.
* Receipt of monoclonal antibody therapy of any kind in the past.
* History of severe reaction to drug infusions or history of severe allergic reactions.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10; Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (2):
- United States (2):
  - The Rockefeller University, New York, New York
  - Weill Cornel Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No pre-assignment phase
Period: Overall Study
Arm/Group | 3BNC117 + ART Interruption
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Adults living with HIV and on suppressive antiretroviral therapy
Arm/Group | 3BNC117 + ART Interruption
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 43 [26 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Rate of Viral Rebound at 12 Weeks After Interruption of Antiretroviral Therapy
Description: Viral rebound is defined as confirmed plasma HIV-1 RNA level > 200 copies/ml in two separate occasions
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 3BNC117 + ART Interruption
Number analyzed (Participants) | 15
Participants | 13

2. Secondary Outcome: Serum Level of 3BNC117 at the Time of Viral Rebound, Measured in Micrograms Per ml
Description: Serum level of 3BNC117 at the time of viral rebound, measured in micrograms per ml
Time Frame: 12 weeks
Population: 3BNC117 serum levels
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | 3BNC117 + ART Interruption
Number analyzed (Participants) | 14
mg/ml | 46.87 (27.67)

3. Secondary Outcome: Time to Viral Rebound After Interruption of Antiretroviral Therapy
Description: Viral rebound is defined as confirmed plasma HIV-1 RNA level > 200 copies/ml in two separate occasions
Time Frame: 36 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | 3BNC117 + ART Interruption
Number analyzed (Participants) | 15
weeks | 5.5 [2 to 17]

4. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Time Frame: 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 3BNC117 + ART Interruption
Number analyzed (Participants) | 17
Participants | 16

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | 3BNC117 + ART Interruption
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3BNC117 + ART Interruption (N=17)
Acute psychotic episode (Psychiatric disorders) | 1 (1) — Hospitalization for an acute psychotic episode 6 days after the second 3BNC117 infusion. Deemed not related to study drug but to underlying bipolar disorder.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3BNC117 + ART Interruption (N=17)
Malaise (General disorders) | 4 (6) — Malaise or fatigue
Nausea (Gastrointestinal disorders) | 4 (4)
Headache (General disorders) | 2 (2)
Dizziness (General disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
This study was an exploratory open label study with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT02588586/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT02588586/ICF_001.pdf